CLINICAL TRIAL: NCT02570035
Title: Protocol for Specified Drug Use-results Survey of Betanis Tablets (for Patients With Coexisting Cardiovascular Disease)
Brief Title: Specified Drug Use-results Survey of Betanis Tablets for Patients With Coexisting Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: BE0003
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Overactive Bladder; Cardiovascular Disease
Keywords: Mirabegron; Overactive Bladder; Cardiovascular Disease
MeSH Terms: conditions — Urinary Bladder, Overactive; Cardiovascular Diseases | interventions — mirabegron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mirabegron group: Subjects with overactive bladder and cardiovascular disease prescribed mirabegron
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — oral
  Other Names: YM178; Betanis

SUMMARY:
This purpose of this study is to investigate the effects of mirabegron on the cardiovascular system in patients with overactive bladder with current or a history of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* having coexisting cardiovascular disease or a history of cardiovascular diseases
* having electrocardiogram record conducted within seven days before the start of the mirabegron treatment (including the first day of administration)

Exclusion Criteria:

* having serious cardiovascular disease
* having significant long QT (QTc > 500 msec)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Overactive bladder patients with current or a history of cardiovascular disease and treated with mirabegron
Sampling Method: Non-Probability Sample
Enrollment: 316 (Actual)
Dates: Start 2012-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Changes in electrocardiogram parameters pre- and post- administration of mirabegron | Baseline and up to four weeks
Incidence rate of cardiovascular system adverse reactions | Up to four weeks
Safety assessed by biochemistry laboratory tests | Up to four weeks
Safety assessed by incidence of adverse events | Up to four weeks

SECONDARY OUTCOMES:
Changes in overactive bladder (OAB) symptoms | Baseline and up to four weeks
  Clinical global impression of change from baseline of OAB symptoms by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (28):
- Japan (28):
  - Site JP81013, Aichi
  - Site JP81014, Aichi
  - Site JP81005, Chiba
  - Site JP81006, Chiba
  - Site JP81007, Chiba
  - Site JP81026, Fukuoka
  - Site JP81027, Fukuoka
  - Site JP81001, Hokkaido
  - Site JP81002, Hokkaido
  - Site JP81021, Hyōgo
  - Site JP81022, Hyōgo
  - Site JP81023, Hyōgo
  - Site JP81024, Hyōgo
  - Site JP81025, Hyōgo
  - Site JP81028, Kagoshima
  - Site JP81011, Kanagawa
  - Site JP81012, Kanagawa
  - Site JP81003, Niigata
  - Site JP81016, Osaka
  - Site JP81017, Osaka
  - Site JP81018, Osaka
  - Site JP81019, Osaka
  - Site JP81020, Osaka
  - Site JP81004, Saitama
  - Site JP81015, Shizuoka
  - Site JP81008, Tokyo
  - Site JP81009, Tokyo
  - Site JP81010, Tokyo